CLINICAL TRIAL: NCT00662077
Title: Study Of The Efficacy And Security Of Ibandronate For Osteoporosis Treatment In A HIV-Infected Patients Cohort
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Financial difficulties
Sponsor: Germans Trias i Pujol Hospital (Other)
Responsible Party: Principal Investigator, Dra. EUGENIA NEGREDO PUIGMAL, Principal Investigator, Germans Trias i Pujol Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VIH-IBAN
Record Dates: First submitted 2008-04-17; First posted 2008-04-21 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: HIV Infections
Keywords: osteoporosis; bifosfonates; ibandronate
MeSH Terms: conditions — HIV Infections; Osteoporosis | interventions — Ibandronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Ibandronate + Lifestyle modifications
  Interventions: Drug: Ibandronate; Behavioral: Lifestyle modifications
- 2 (Other): Lifestyle modifications
  Interventions: Behavioral: Lifestyle modifications

INTERVENTIONS:
Drug: Ibandronate — Ibandronate endovenous 3 mg every 3 months
  Arms: 1
Behavioral: Lifestyle modifications — Lifestyle modifications: counseling every 3 months

SUMMARY:
This project wills to determine the incidence of osteoporosis in our population of HIV-infected patients and to assess the efficacy and security of ibandronate, whose efficacy in post-menopausal women has already been proved.

DETAILED DESCRIPTION:
The lower bone mineral density that has been described in patients with HIV-infection has not meant an increase of long term complications. Nevertheless, it could involve an increase if the associated co-mordibity in the future, taking in care that in general population osteoporosis increases 4 times the pathologic fracture risk. That's why it is necessary to know the real prevalence of osteoporosis in this population of patients so the real dimensions of the problems can be defined.

This project wills to determine the incidence of osteoporosis in our population of HIV-infected patients and to assess the efficacy and security of ibandronate, whose efficacy in post-menopausal women has been already proved. If the quarterly use of endovenous ibandronate obtains equivalent results to those obtained with oral and weekly alendronate in other studies with the same population, its use would be justified because of its posology benefits. The monthly or quarterly administration can improve compliance in patients who are recieving a big quantity of drugs, as HIV infected patients do and who probably have to be treated for life. Moreover, its elimination is renal so there is absence of interactions with antiretroviral drugs what mades of ibandronate a very promising alternative. Finally, there's no risk of digestive intolerance because of its parenteral administration and it has a better posology than oral bifosfonates.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old or elder.
2. Documented HIV-1 infection, with or without antiretroviral treatment.
3. Presence of WHO osteoporosis criteria, defined as t-score under -2.5 in lumbar, hip and/or trochanter. (DEXA in the last 6 months is needed)
4. Willing to follow the study protocol.
5. Informed Consent signature.

Exclusion Criteria:

1. In women, pregnancy or breastfeeding.
2. Other possible causes of secondary osteoporosis.
3. Creatinin over 2.3mg/mL
4. Glomerular filter less than 50 mL/min (estimated through MDRD)
5. Alendronate treatment in the last 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Increase in lumbar (L2-4) and femoral (trochanter, femur neck, total femur and hip) t-score bone mineral density | BL, W24, W48, W72, W96

SECONDARY OUTCOMES:
Adverse events | BL, W12, W24, W36, W48, W60, W72, W80, W96
Lab tests | BL, W12, W24, W36, W48, W60, W72, W80, W96
Related clinical events (bone fractures) | BL, W12, W24, W36, W48, W60, W72, W80, W96
Osteoblastic/Osteoclastic activity, bone formation/reabsorption. | BL, W12, W24, W36, W48, W60, W72, W80, W96

CONTACTS AND LOCATIONS:
Overall Officials: Eugenia Negredo, MD,PhD, Principal Investigator — Fundación FLS de Lucha Contra el Sida, las Enfermedades Infecciosas y la Promoción de la Salud y la Ciencia
Locations (1):
- Germans Trias i Pujol Hospital - Lluita Sida Foundation, Badalona, Barcelona, Spain